CLINICAL TRIAL: NCT00471887
Title: A Phase II, Open-Label, Single Arm Clinical Trial to Study the Mechanism of Action of CP-675,206 in Patients With In-Transit and Metastatic Melanoma Amenable to Repeated Outpatient Tumor Biopsies
Brief Title: Ticilimumab (CP-675,206) in Treating Patients With Stage IIIC or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-0002360; UCLA-0606093-01; PFIZER-UCLA-0606093-01; CDR0000543416 (Other: UCLA IRB)
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2016-01

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment-Single Arm (Experimental): See intervention descriptions
  Interventions: Biological: CP-675,206

INTERVENTIONS:
Biological: CP-675,206 — Patients will receive intravenous administration of CP-675,206 at a dose of 15mg/kg on Day 1 of an every 90 day cycles. For purposes of treatment visits and scheduling, each cycle is defined as a 90 day period. Patients may receive up to 8 dose (8 cycles) in a 24-month period until progression of disease or intolerable toxicity.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as ticilimumab (CP-675,206), can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase II trial is studying how well ticilimumab (CP-675,206) works in treating patients with stage IIIC or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the change in melanoma intratumoral infiltrates by cluster of differentiation 8 (CD8 positive) cytotoxic T lymphocytes in patients with stage IIIC or IV melanoma treated with ticilimumab (CP-675,206).

Secondary

* Determine the effects of this drug on intratumoral immune effector cells and tumor cells in these patients.
* Determine the effects of this drug on circulating immune effector cells in these patients.
* Determine the gene expression profile of immune effector cells and tumor cells in regressing and nonregressing tumors in these patients.
* Bank plasma from peripheral blood obtained from patients with regressing and nonregressing tumors for future exploratory analysis of proteomic profile.
* Assess additional evidence of antitumor activity of this drug, as measured by best on-study response rate, in these patients.
* Characterize the safety profile and tolerability of this drug in these patients.
* Obtain pharmacokinetic data to be used in a future meta-analysis of this drug's pharmacokinetics.
* Determine whether the CTLA4 genotype influences the safety, immune response, and/or efficacy of this drug in these patients.
* Determine the relationships between clinical response (i.e., efficacy or toxicity) and tumor and/or blood ex vivo analysis in patients treated with this drug.

OUTLINE: This is an open-label, randomized study.

Patients receive ticilimumab (CP-675,206) IV over 2 hours on day 1. Treatment repeats every 90 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection periodically during study for correlative pharmacokinetic (PK), pharmacogenetic, and pharmacogenomic analyses. Blood specimens are obtained for PK measurement at baseline and periodically during study treatment for analysis by enzyme-linked immunosorbent assay. Blood specimens are also evaluated by pharmacogenetic assessment of polymorphisms in CTLA4. Patients also undergo leukapheresis at baseline and at least once between days 30-60 for biomarker analysis of immune cell activation (i.e.,biomarkers CD45RO, CD45RA, HLA-DR, CCR5, CCR7, CD62L, CD69); Treg phenotype (i.e., CD4/CD25/GITR/intracellular FoxP3); and Treg function. In HLA-A2.1 positive patients, peripheral blood mononuclear cells (PBMC) are analyzed for antigen-specific immune reactivity by MART-1, gp100, and tyrosine MHC tetramer using enzyme-linked immunosorbent spot assay. Plasma obtained during leukapheresis is assessed for levels of circulating cytokines and chemokines. Some plasma is stored for future proteomic profile analysis.

Patients also undergo excisional or punch biopsy at baseline and between days 30-60 during course 1. Tumor tissue samples embedded in paraffin are analyzed by hematoxylin-eosin and immunohistochemical staining for several biomarkers, including biomarkers of immune cell response (i.e., cluster of differentiation 3 (CD3), cluster of differentiation 4 (CD4), and cluster of differentiation 8 (CD8) and biomarkers of melanoma (i.e., S-100, MART-1, and/or HMB45). Frozen tumor tissue samples are analyzed by gene chips and gene arrays for gene expression profile and by quantitative real-time polymerase chain reaction for FoxP3. Minced tumor tissue samples are analyzed by flow cytometry in nonadherent cells for HLA-DR (if tumor-infiltrating lymphocytes are available) and by Braf sequencing in adherent cells (if melanoma cells are available).

After completion of study therapy, patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 21 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma that is surgically incurable and either:

  * Stage IIIc melanoma including locally relapsed, satellite, in-transit lesions or bulky draining lymph node metastasis.
  * Stage IV melanoma (M1a, M1b, M1c) with accessible lesions for biopsy.
* At least 2 lesions amenable for outpatient biopsies
* No restriction based on prior treatments
* Disease progression after the last dose of prior therapy
* A minimum of one measurable lesion defined as:

  * Meeting the criteria for measurable disease according to Response Evaluation Criteria in Solid Tumors
  * Skin lesion(s) selected as non-completely biopsied target lesions that can be accurately measured and recorded by color photography with a ruler to document the size of the target lesion(s).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate bone marrow and hepatic function determined within 30 days prior to enrollment, defined as:

  * Absolute neutrophil count > 1.0 x 10^9 cells/L
  * Platelets > 90 x 10^9 /L
  * Hemoglobin > 9 g/L
  * Aspartate and alanine aminotransferases < 2.5 x upper limit of normal (ULN) (< 5 x ULN, if documented liver metastases are present)
  * Total bilirubin < 2 x ULN (except patients with documented Gilbert's syndrome)
* Must be willing and able to provide writing informed consent.
* Must be willing and able to accept at least two tumor biopsies.
* Must be willing and able to accept at least two leukapheresis procedures.

Exclusion Criteria:

* Received treatment for cancer, including immunotherapy, within one month prior to dosing.
* Previous participation in Pfizer study A3671009: A Phase 3, Open Label, Randomized Comparative Study of CP-675,206 and Either Dacarbazine or Temozolomide in Patients with Advanced Melanoma
* Eligible for enrollment to Pfizer A3671008: A Phase 2, Open Label, Single Arm Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of CP-675,206 in Patients with Advanced Refractory and/or Relapsed Melanoma
* History of significant evidence of risk for chronic inflammatory or autoimmune disease. Patents will be eligible if prior autoimmune disease of the hypophysis was treated locally or have resulted in fibrotic damage requiring thyroid hormone replacement. Vitiligo will not be a basis for exclusion.
* History of inflammatory bowel disease, celiac disease, or other chronic gastrointestinal conditions associated with diarrhea or bleeding, or current acute colitis or any origin
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 4 weeks prior to enrollment
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
* Clinically active brain metastases. Radiological documentation of absence of brain metastases at screening is required for all patients
* Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01; Primary Completion 2011-07 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, MD, Principal Investigator — Jonsson Comprehensive Cancer Center; John A. Glaspy, MD, MPH, Principal Investigator — Jonsson Comprehensive Cancer Center; James S. Economou, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Background] von Euw E, Chodon T, Attar N, Jalil J, Koya RC, Comin-Anduix B, Ribas A. CTLA4 blockade increases Th17 cells in patients with metastatic melanoma. J Transl Med. 2009 May 20;7:35. doi: 10.1186/1479-5876-7-35. PMID 19457253
- [Derived] Huang RR, Jalil J, Economou JS, Chmielowski B, Koya RC, Mok S, Sazegar H, Seja E, Villanueva A, Gomez-Navarro J, Glaspy JA, Cochran AJ, Ribas A. CTLA4 blockade induces frequent tumor infiltration by activated lymphocytes regardless of clinical responses in humans. Clin Cancer Res. 2011 Jun 15;17(12):4101-9. doi: 10.1158/1078-0432.CCR-11-0407. Epub 2011 May 10. PMID 21558401
- [Derived] Comin-Anduix B, Sazegar H, Chodon T, Matsunaga D, Jalil J, von Euw E, Escuin-Ordinas H, Balderas R, Chmielowski B, Gomez-Navarro J, Koya RC, Ribas A. Modulation of cell signaling networks after CTLA4 blockade in patients with metastatic melanoma. PLoS One. 2010 Sep 15;5(9):e12711. doi: 10.1371/journal.pone.0012711. PMID 20856802

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: CP-675,206 Monoclonal Antibody.: See intervention descriptions
  CP-675,206: Patients will receive intravenous administration of CP-675,206 at a dose of 15mg/kg on Day 1 of an every 90 day cycles. For purposes of treatment visits and scheduling, each cycle is defined as a 90 day period. Patients may receive up to 8 dose (8 cycles) in a 24-month period until progression of disease or intolerable toxicity.
Period: Overall Study
Arm/Group | Treatment: CP-675,206 Monoclonal Antibody.
Started | 32
Completed | 23
Not Completed | 9
Not completed — Adverse Event | 9

BASELINE CHARACTERISTICS:
Arm/Group | Treatment: CP-675,206 Monoclonal Antibody
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: years] | 52 [27 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 32
prior therapies [Number; unit: participants]
  No Prior Therapy | 13
  Biological Only | 4
  Chemotherapy Based | 13
  Other | 2
Stage [Number; unit: participants] — American Joint Committee on Cancer Melanoma of the Skin Staging for disease staging.
  IIIc: Tumor thickness, no detectable evidence of distant metastases M1a: metastases to skin M1b: Metastases to lung M1c: Metastases to all other visceral sites or distant metastases The progression is M1a, M1b and M1c with M1c being worse. Scan results were used to confirm melanoma stage of patients. For Stage IIIc the scans showed melanoma spread to the lymph nodes and for Stage IV melanoma metastasized distant skin/soft tissue (M1a), lung (M1b) or other location excluding central nervous system (M1c).
  participants
    IIIC | 4
    M1a | 3
    M1b | 3
    M1c | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor Infiltration by Cluster of Differentiation 8 (CD8) Positive Cytotoxic T Lymphocytes
Description: Tumor infiltration of cluster of differentiation 4 and cluster of differentiation 8 (CD4+ and CD8+) cells (intratumoral and peritumoral) was assessed by immunohistochemistry of tumor tissue obtained through biopsy before and after administration of tremelimumab. Up to 10 randomly selected fields per sample were analyzed.
Time Frame: pre treatment - post treatment at 24 months
Population: 19 (4 Responders and 15 Non-responders) Outcome data summary: An increase in intratumoral infiltration of lymphocytes following administration of tremelimumab independent of clinical response is expected
Measure: Mean (Standard Error); unit: cells/mL
Arm/Group | Treatment: CP-675,206 Monoclonal Antibody
Number analyzed (Participants) | 19
cells/mL
  Pre-Treatment (cell density)Intratumoral CD8+ | 289 (61)
  Pre-Treatment (cell density)Intratumoral CD4+ | 104 (32)
  Post-Treatment (cell density)Intratumoral CD8+ | 955 (191)
  Post-Treatment (cell density)Intratumoral CD4+ | 428 (156)

2. Secondary Outcome: Change in Intratumoral Expression of the Proteins HLA-DR, CD45RO, Ki67 and FOXP3 and FOXP3"
Description: HLA-DR is a surface marker of T cell activation after exposure to CTLA4 blocking antibodies. CD45RO is a maker of prior cognate antigen-exposed T cells. Together they mark cells with a surface phenotype of T effector or T effector memory cells. Ki67 is a marker of cell proliferation. The protein FOXP3 is involved in the regulation of the development and function of regulatory T cells, and serves as a marker of this cell type. Intratumoral expression of HLA-DR, CD45RO, Ki67 and FOXP3 was assessed by immunohistochemistry of tumor tissue obtained through biopsy before and after administration of tremelimumab.
Time Frame: pre treatment - post treatment at 24 months
Population: 11 (3 Responders and 8 Non-responders)
Measure: Mean (Standard Deviation); unit: cells/mL
Arm/Group | Treatment: CP-675,206 Monoclonal Antibody
Number analyzed (Participants) | 11
cells/mL
  HLA-DR/CD45RO | 356.4 (257.33)
  Ki67 | -240.26 (690.48)
  FOXP3 | 132.15 (160.35)

3. Secondary Outcome: Differences in Morphological and Gene Expression Profiling Studies in Peripheral Blood Mononuclear Cells
Description: T cell receptor (TCR) usage was analyzed in genomic DNA from peripheral blood from patients before and after treatment with tremelimumab. High-throughput deep sequencing of the TCR Vβ CDR3 (Complementarity - determining region 3) region was analyzed to better characterize the expansion and clonality of the T cell repertoire.
  The frequency of circulating invariant natural killer T cells (iNKT) cell subsets were also characterized by flow cytometry in peripheral blood samples pre- and post-treatment. iNKT cells regulate the balance of Th1/Th2 immune responses.
Time Frame: pre treatment - post treatment at 24 months
Population: 21 (4 Responders and 17 Non-responders)
Measure: Mean (Standard Deviation); unit: cell density (number of cells/mm^2)
Arm/Group | Treatment: CP-675,206 Monoclonal Antibody
Number analyzed (Participants) | 21
cell density (number of cells/mm^2)
  CD4+iNKT pre-treatment | 104 (32)
  CD4+iNKT post-treatment | 428 (156)

4. Secondary Outcome: Changes in the Protein Content in Peripheral Blood With an Increase in Proinflammatory Cytokines and Chemokines
Description: Th17 cells are CD4+ cells that are potent inducers of tissue inflammation and autoimmunity. The levels of this T cell subset were assessed in peripheral blood from patients before and after administration of tremelimumab. Th17 cells were assessed since the major dose limiting toxicities are inflammatory and autoimmune in nature.
  In addition, the phosphorylation of signaling molecules downstream of the TCR and cytokine receptors was evaluated in peripheral blood cells from patients before and after treatment with tremelimumab using intracellular flow cytometry.
  ab#cells = absolute number of cells
Time Frame: pre treatment - post treatment at 24 months
Population: 21 (4 Responders and 17 Non-responders)
Measure: Median (95% Confidence Interval); unit: absolute number of cells
Arm/Group | Treatment: CP-675,206 Monoclonal Antibody
Number analyzed (Participants) | 21
absolute number of cells
  Peripheral Blood Pre-treatment: pg/ml x 1E6cells | 73711 [46912 to 100510]
  Peripheral Blood Post-treatment: pg/ml x 1E6cells | 101066 [70644 to 131488]
  Unstimulated CD4+Pre-Treatment | 0.46 [0.22 to 0.7]
  Unstimulated CD4+Post-Treatment | 0.62 [0.49 to 0.75]

5. Secondary Outcome: Overall Response (Complete or Partial Response) as Measured by RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression
Time Frame: pre treatment - post treatment at 24 months
Measure: Number; unit: participants
Arm/Group | Treatment: CP-675,206 Monoclonal Antibody
Number analyzed (Participants) | 31
participants
  Progressive Disease | 27
  Partial Response | 1
  Complete Response | 3

6. Secondary Outcome: Overall Safety Profile as Measured by NCI CTCAE v2.0
Time Frame: pre treatment - post treatment at 24 months
Measure: Number; unit: participants
Arm/Group | Treatment: CP-675,206 Monoclonal Antibody
Number analyzed (Participants) | 32
participants
  Seroius Adverse Event (SAE)SAE | 13
  Adverse Events (AE) | 13

ADVERSE EVENTS:
Time Frame: From time of consent until 30 after last treatment. Up to 1 year.
Groups:
- Treatment-CP-675,206: See intervention descriptions
  CP-675,206: Patients will receive intravenous administration of CP-675,206 at a dose of 15mg/kg on Day 1 of an every 90 day cycles. For purposes of treatment visits and scheduling, each cycle is defined as a 90 day period. Patients may receive up to 8 dose (8 cycles) in a 24-month period until progression of disease or intolerable toxicity.
Arm/Group | Treatment-CP-675,206
All-Cause Mortality (participants affected / at risk) | 13/32
Serious Adverse Events (participants affected / at risk) | 13/32
Other Adverse Events (participants affected / at risk) | 13/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-CP-675,206 (N=32)
Chronic Immune Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 9 (9)
Pruritius (Skin and subcutaneous tissue disorders) | 3 (3)
Hypophysitis (Immune system disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-CP-675,206 (N=32)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
dyspena (Respiratory, thoracic and mediastinal disorders) | 4 (4)
hypotension (Cardiac disorders) | 1 (1)
tumor pain (General disorders) | 1 (1)
tachycardia (Cardiac disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 6 (6)
ertherma biopsy site (General disorders) | 1 (1)
bronchitis (Infections and infestations) | 1 (1)
fever (Infections and infestations) | 3 (3)
pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
nausea (General disorders) | 3 (3)
insomnia (General disorders) | 1 (1)
itchness (General disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 4 (4)
loss of right eye vision (Eye disorders) | 1 (1)
lower back pain (General disorders) | 2 (2)
nocturia (Renal and urinary disorders) | 1 (1)
sleepiness (General disorders) | 2 (2)
night sweats (General disorders) | 1 (1)
neck pain (General disorders) | 1 (1)
anemia (General disorders) | 2 (2)
fatigue (General disorders) | 1 (1)
asthenia (General disorders) | 1 (1)
headaches (General disorders) | 1 (1)
right hip pain (General disorders) | 1 (1)
colitis (Gastrointestinal disorders) | 2 (2)
abdominal pain (General disorders) | 2 (2)
weight loss (General disorders) | 1 (1)
acute renal failure (Renal and urinary disorders) | 1 (1)
dizziness (General disorders) | 1 (1)
depression (General disorders) | 1 (1)
anxiety (General disorders) | 1 (1)
cold (Infections and infestations) | 1 (1)
diplopia (Eye disorders) | 1 (1)
hypophysitis (Blood and lymphatic system disorders) | 1 (1)
leg twitiching (General disorders) | 1 (1)
perforated colon (Gastrointestinal disorders) | 1 (1)
left side pain (General disorders) | 1 (1)
brain metastasis (Nervous system disorders) | 1 (1)
left nares maxilla swelling (General disorders) | 1 (1)
left nares maxilla bleeding (General disorders) | 1 (1)
shortness of breath (General disorders) | 1 (1)
bleeding lesion (General disorders) | 1 (1)
confusion (General disorders) | 1 (1)
oozing from bulky right axillary mass (General disorders) | 1 (1)
groves disease (Skin and subcutaneous tissue disorders) | 1 (1)
edema left low extremity (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No